CLINICAL TRIAL: NCT04310111
Title: Efficacy and Safety of Endoscopic Ultrasonography-guided Radiofrequency Ablation in Treatment of Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: EUS-RFA for Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Associate director of gastroenterology department, First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-01-112
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic ductal adenocarcinoma; Unresectable pancreatic cancer; Radiofrequency ablation; Endoscopic ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-RFA (Experimental): Patients were placed in the lateral position under deep sedation with supplementary oxygen and electrocardiograph monitoring. The target tumor was identified by EUS, then the biopsy needle stylet was removed and replace with the RFA probe. RF energy was applied for 90-120 seconds at 5 Watts. Wait 1 minute before repositioning the Habib™ EUS RFA needle and repeat procedure as many times as needed to ensure complete ablation of the tumor. EUS-guided celiac plexus neurolysis (EUS-CPN) was performed on patients with intractable upper abdominal pain.
  Interventions: Procedure: EUS-RFA

INTERVENTIONS:
Procedure: EUS-RFA — Use EUS-RFA to treat unresectable pancreatic cancer

SUMMARY:
The clinical application of intraoperative or percutaneous radiofrequency ablation (RFA) for pancreatic ductal adenocarcinoma (PDAC) is limited due to higher mortality and incidence of adverse events. The aim of this study was to evaluate the efficacy and safety of endoscopic ultrasonography-guided RFA (EUS-RFA) for locally advanced, unresectable PDAC. Patients with unresectable PDAC who underwent EUS-RFA were included from September 2013 to June 2016. Pre- and post-procedural clinical data was retrospective collected.

DETAILED DESCRIPTION:
evaluate the efficacy and safety of endoscopic ultrasonography-guided RFA (EUS-RFA) for locally advanced, unresectable PDAC.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 80 years old. ② unresectable PDAC based on review of abdominal cross-sectional imaging (CT or MRI) and cytology/ histology results. ③Intolerance to chemotherapy due to side effects or patient's comorbidities.

Exclusion Criteria:

* Pregnancy or breast-feeding；②ECOG performance status 3 or 4；③Patients with distant metastases or malignant ascites, life expectancy less than 3 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Tumor size | 2 years
  Tumor size

SECONDARY OUTCOMES:
Serum levels of CA19-9 | 2 years
  Serum levels of CA19-9 before and after surgery
survival rate | 2 years
  including Overall survival
Adverse events | 2 years
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No